CLINICAL TRIAL: NCT06609928
Title: A Phase 1 Study of FOLR1 CAR T for Pediatric Patients With FOLR1/CBFA2T3::GLIS2+ Relapsed or Refractory AML
Brief Title: FH-FOLR1 Chimeric Antigen Receptor T Cell Therapy for Treating Pediatric Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Kuni Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1124385; NCI-2024-06808 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00004888 (Other: Fred Hutch/University of Washington/Seattle Children's Cancer Consortium)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Childhood Acute Myeloid Leukemia; Refractory Childhood Acute Myeloid Leukemia
MeSH Terms: interventions — Specimen Handling; Biopsy; Cyclophosphamide; fludarabine; Blood Component Removal; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (FH-FOLR1 CAR T) (Experimental): Patients undergo apheresis to obtain T cells for product manufacturing. Patients receive lymphodepleting chemotherapy with fludarabine IV on days -4 to -1 and cyclophosphamide IV on days -4 and -3. Patients receive FH-FOLR1 CAR T IV on day 0. Patients undergo ECHO at screening, undergo collection of CSF and blood samples and bone marrow aspiration/biopsy throughout the study, and may undergo PET scan on study and during follow up.
  Interventions: Biological: FOLR1 CAR T-cells; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cyclophosphamide; Procedure: Echocardiography Test; Drug: Fludarabine; Procedure: Pheresis; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: FOLR1 CAR T-cells — Given IV
  Other Names: Anti-FOLR1 CAR-T Cells; FH-FOLR1 CAR T Cells
Procedure: Biospecimen Collection — Undergo CSF and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Pheresis — Undergo apheresis
  Other Names: Apheresed; Apheresis; Blood Component Removal; Collection, Apheresis/Leukapheresis; Hemapheresis
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of FH-FOLR1 chimeric antigen receptor (CAR) T cells in treating pediatric patients with FOLR1+ acute myeloid leukemia (AML) that has come back after a period of improvement (recurrent) or has not responded to previous treatment (refractory). CAR T-cell therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a FOLR1 on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor. Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Chemotherapy drugs, such as fludarabine and cyclophosphamide, are given to a patient before the manufactured FH-FOLR1 CAR T cells are infused back into the patient to assist in the CAR T cell activity in the patient. The trial is evaluating if giving FH-FOLR1 CAR T cell therapy is safe and tolerable for pediatric patients with recurrent or refractory AML.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of FH-FOLR1 CAR T.

Patients undergo apheresis to obtain T cells for product manufacturing, receive lymphodepleting chemotherapy with fludarabine intravenously (IV) on days -4 to -1, cyclophosphamide IV on days -4 and -3 and receive FH-FOLR1 CAR T IV on day 0. Patients undergo echocardiography (ECHO) at screening, undergo collection of cerebrospinal fluid (CSF), blood samples and bone marrow aspiration/biopsy throughout the study, and may undergo imaging (such as positron emission tomography (PET) scan).

After completion of study treatment, patients are followed up for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject age ≤ 6 years.
* Weight ≥ 7 kilograms.
* AML that expresses FOLR1 by flow cytometry as assessed by Hematologics, Inc.

Laboratory and meets one of the below definitions:

* For subjects who have previously received an allogeneic hematopoietic cell transplantation (HCT), any evidence of AML re-emergence post HCT detectable by flow cytometry.
* First relapse of AML ≤ 6 months from initial diagnosis.
* First relapse of AML > 6 months from initial diagnosis with minimal residual disease (MRD) ≥ 0.05% by flow cytometry after at least one re-induction attempt (one cycle of therapy).
* Second or greater relapse of AML.
* Refractory AML, defined as ≥ 0.1% leukemic cells determined by flow cytometry or > 1% on biopsy after 2 cycles of chemotherapy.

  * Able to tolerate apheresis.
  * Life expectancy ≥ 8 weeks.
  * Has an appropriate stem cell donor source identified.
  * Lansky performance status score of ≥ 50. Subjects who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for purposes of assessing performance status.
  * The subject must discontinue all anticancer agents and radiotherapy and, in the opinion of the investigator, have fully recovered from significant acute toxic effects of all prior chemotherapy, immunotherapy, and radiotherapy:
* Chemotherapy and biologic agents: All chemotherapy and biologic therapy not specifically mentioned below must be discontinued ≥ 14 days prior to enrollment, with the exception of intrathecal chemotherapy for which there is not a required washout period.
* Steroid use: All corticosteroid therapy (unless physiologic replacement dosing) must be discontinued ≥ 7 days prior to enrollment, unless being used to treat graft-versus-host disease (GVHD) (if being used to treat GVHD see requirements).
* Tyrosine kinase inhibitor (TKI) use: All TKIs must be discontinued ≥ 3 days prior to enrollment.
* Hydroxyurea: must be discontinued ≥ 1 day prior to enrollment.
* FOLR1 targeting therapy must be discontinued within 30 days prior to enrollment.

  * Gene modified cellular therapy:
* Must be at least 30 days from most recent gene modified cell therapy infusion and document no evidence of modified cells in the peripheral blood OR
* Must be at least 60 days from most recent gene modified cell therapy.

  * Serum creatinine ≤ 1.5 x the upper limit of normal (ULN) based on the following:
* Age 1 to < 2 years: maximum serum creatinine 0.6 mg/dL for male and 0.6 mg/dL for female.
* Age 2 to < 6 years: maximum serum creatinine 0.8 mg/dL for male and 0.8 mg/dL for female.
* Age 6 to < 10 years: maximum serum creatinine 1 mg/dL for male and 1 mg/dL for female.

  * Total bilirubin ≤ 3 times ULN for age OR conjugated bilirubin ≤ 2 mg/dL.
  * Alanine aminotransferase (ALT)(serum glutamic-pyruvic transaminase [SGPT]) ≤ 5 times ULN.
  * Shortening fraction ≥ 28% OR ejection fraction (EF) ≥ 50% as measured by echocardiogram.
  * Oxygen saturation ≥ 92% on room air without supplemental oxygen or mechanical ventilation.
  * Absolute lymphocyte count (ALC) ≥ 100 cells/uL.
  * Virology testing negative within 3 months prior to enrollment, to include:
* HIV antigen & antibody.
* Hepatitis B surface antigen.
* Hepatitis C antibody OR if positive, hepatitis C polymerase chain reaction (PCR) is negative.

  * Subject and/or legally authorized representative has signed the informed consent form for this study.

Exclusion Criteria:

* Active malignancy other than acute myeloid leukemia.
* History of symptomatic non-AML central nervous system (CNS) disease or ongoing symptomatic CNS disease requiring medical intervention, including paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injury, dementia, cerebellar disease, organic brain syndrome, psychosis, coordination or movement disorder (subjects with non-febrile seizure disorder controlled on anti-epileptic medication and without seizure activity within 1 month are eligible).
* CNS AML involvement that is symptomatic and in the opinion of the investigator, cannot be controlled during the interval between enrollment and T cell infusion.
* If history of allogeneic stem cell transplant: active GVHD or receiving immunosuppressive therapy for treatment or prevention of GVHD within 4 weeks prior to enrollment.
* If history of allogeneic stem cell transplant and patient has received donor lymphocyte infusion (DLI) the subject is < 8 weeks from DLI infusion.
* Presence of active severe infection, defined as:

  * Positive blood culture within 48 hours of enrollment, OR
  * Fever above 38.2 degrees Celsius (C), AND clinical signs of infection within 48 hours of enrollment.
* Primary immunodeficiency syndrome.
* Subject has received prior virotherapy.
* Subject and/or legally authorized representative unwilling to provide consent/assent for participation in the 15-year follow-up period, required if FH-FOLR1 CAR T cell therapy is administered.
* Presence of any condition that, in the opinion of the investigator, would prohibit the subject from undergoing treatment under this protocol.
* Considered by the investigator to be unable to tolerate a lymphodepleting regimen.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2042-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 15 years
  Will be summarized in terms of type, severity, date of onset, and attribution using the Common Terminology for Adverse Events version 5.
Rate of manufacturing anti-FOLR1 chimeric antigen receptor (CAR) T-cells (FH-FOLR1 CAR T) product | Up to 28 days
  Feasibility will be determined by the rate of manufacturing a FH-FOLR1 CAR T cell product from apheresis product.

SECONDARY OUTCOMES:
Aplasia | At 42 days
  Will be defined as if a patient has a hypoplastic bone marrow and has failure to recover a peripheral absolute neutrophil count > 200/uL and a non-transfusion dependent platelet count > 20,000/uL not due to malignant infiltration or severe infection (defined as ≥ grade 3 infection). Will be assessed using peripheral blood and bone marrow.
Persistence of FH-FOLR1 CAR T | Up to 15 years
  FOLR1 persistence will be defined as detection of the FH-FOLR1 CAR T by flow or polymerase chain reaction above the lower limit of detection. Will be assessed by peripheral blood.
Overall survival | From infusion of FH-FOLR1 CAR T cell product to death from any cause, assessed up to 15 years
Disease free survival | From T cell infusion to the first observation of disease or death fromany cause, whichever occurs first, assessed up to 15 years
Duration of overall response | From the time criteria are met for complete response or partial response until the first date that treatment failure is objectively documented, assessed up to 15 years
Non-relapse mortality | From T cell infusion to death where cause of death is not attributable tounderlying disease, assessed up to 15 years
Event free survival | From infusion of FH-FOLR1 CAR T product to an event, with eventsdefined as relapse, secondary malignancy, death from any cause, assessed up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Katherine G. Tarlock, MD, Principal Investigator — Fred Hutch/University of Washington/Seattle Children's Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington/Seattle Children's Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No